CLINICAL TRIAL: NCT05166655
Title: Intra-operative Recordings to Characterize Movement Facilitation in Parkinson's Disease
Brief Title: DBS Recordings to Characterize Movement Facilitation in Parkinson's Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kathryn A. Cross, MD, PhD, Assistant Professor in Residence, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-001271; 1K23NS119568 (NIH)
Record Dates: First submitted 2021-12-16; First posted 2021-12-22 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: deep brain stimulation; neuromodulation; external cueing; movement
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parkinson disease patients (Experimental): Parkinson disease patients undergoing DBS Surgery of the Globus Pallidus Internus (GPi) for clinical indications
  Interventions: Behavioral: Movement task

INTERVENTIONS:
Behavioral: Movement task — Computer task with experimental conditions manipulating sensory and motivation cues for movement.

SUMMARY:
Several strategies or contexts help patients with Parkinson's disease to move more quickly or normally, however the brain mechanisms underlying these phenomena are poorly understood. The proposed studies use intraoperative recordings during DBS surgery for Parkinson's disease to understand the brain mechanisms supporting improved movements elicited by external cues. The central hypothesis is that distinct networks are involved in movement improvement depending on characteristics of the facilitating stimulus. Participants will perform movement tasks during awake surgery performed exclusively for clinical indications. The identified biomarkers may provide targets for future neuromodulation therapies to improve symptoms that are refractory to current treatments, such as freezing of gait.

DETAILED DESCRIPTION:
Patients with Parkinson's disease (PD) will perform computer tasks involving reaching and tapping movements during video recording of movements and electrophysiological recording of brain signals during deep brain stimulation surgery. Experimental manipulations involve different computer stimuli that manipulate the presence or absence of sensory and motivational movement cues. The same experimental manipulations are delivered to all individual subjects. 40 PD patients who are undergoing deep brain stimulation (DBS) surgery for treatment of Parkinson's disease, will perform the tasks during awake surgery and recordings will be obtained from 2 implanted DBS electrodes as well as 2 temporary electrode strips placed on the surface of the brain for research purposes. Study procedures are limited to the intraoperative environment with no additional study visits. All patients will also be asked to perform clinical rating scales and questionnaires and undergo a movement disorders neurological exam.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease based on presence of at least 2 cardinal PD features (tremor, rigidity, or bradykinesia)
* Undergoing deep brain stimulation surgery for treatment of advanced Parkinson's disease, according to clinical evaluation, including the following criteria:
* advanced idiopathic PD as determined by OFF unified Parkinson's Disease Rating Scale (UPDRS) part III motor subscale > 25
* L-dopa responsive symptoms with at least 30% improvement in UPDRS III scores on vs. off medication OR medication refractory disabling tremor
* Persistent disabling motor symptoms or drug side effects (dyskinesias, motor fluctuations, disabling "off" periods) despite optimal medical therapy
* preoperative MRI without evidence of cortical or subdural adhesions or vascular abnormalities
* Willingness and ability to cooperate during conscious operative procedure for up to 40 minutes

Exclusion Criteria:

* medical contraindication to surgery, including use of anticoagulant or antiplatelet therapy within 1 week
* significant cognitive or psychiatric disease based on clinical neuropsychological testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Globus pallidus internus local field potentials | baseline
  power in the beta band
Frontal and parietal electrocorticography | baseline
  power in the beta band

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Electrophysiological and behavioral data obtained during task performance will be made available upon request to Dr. Cross (PI) via secured server access. Data sharing agreement will be required for all requests.